CLINICAL TRIAL: NCT00532766
Title: Bioequivalence of Jusline Following Subcutaneous Administration in Healthy Subjects
Brief Title: Evaluating Pharmacokinetics and Pharmacodynamics of Jusline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRC06-535
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Healthy
Keywords: Healthy subjects
MeSH Terms: interventions — Insulin, Regular, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Experimental): Jusline Humulin
  Interventions: Drug: Jusline

INTERVENTIONS:
Drug: Jusline
  Other Names: Humulin

SUMMARY:
To evaluate the pharmacokinetic and pharmacodynamic profile of a new human insulin (Jusline) after subcutaneous administration, and to compare this profile with Humulin insulin.

DETAILED DESCRIPTION:
To study the pharmacokinetic and pharmacodynamic profile of a new human insulin (Jusline) after subcutaneous administration in the abdominal, and to compare this profile with Humulin insulin for three different preparations (Regular, NPH, and Premixed Regular/NPH (30/70)).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-diabetic
* Age 18-35 year
* Normal body mass index (BMI 18-25 kg/m2)

Exclusion Criteria:

* Diabetics
* Overweight/obese
* Anemic, with liver, cardiac, renal or thyroid dysfunction

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic and pharmacodynamic profile of a new human insulin (Jusline)

CONTACTS AND LOCATIONS:
Overall Officials: Khalid A Al-Rubeaan, MD, Principal Investigator — College of Medicine, King Saud University
Locations (1):
- University Diabetes Center, Riyadh, Riyadh Region, Saudi Arabia